CLINICAL TRIAL: NCT02920450
Title: A Non-Randomized Phase Ib-II Protocol of Paclitaxel, Carboplatin and the Dual PI3K/mTOR Kinase Inhibitor, PF-05212384, for Patients With Advanced, or Metastatic Non-Small Cell Carcinoma of the Lung
Brief Title: Study of Paclitaxel, Carboplatin, and PF-05212384 in Advanced or Metastatic NSCLC (UF-STO-LUNG-002)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Florida (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601181 -A; WI211924 (Other: Pfizer Inc.); UF-STO-LUNG-002 (Other: University of Florida); OCR15075 (Other: University of Florida)
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: lung; carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — gedatolisib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Arm (Phase 1b; Gedatolisib Dose Level 1[110 mg]) (Experimental)
  Interventions: Drug: Gedatolisib; Drug: Paclitaxel; Drug: Carboplatin
- Treatment Arm (Phase 1b; Gedatolisib Dose Level 2[150 mg]) (Experimental)
  Interventions: Drug: Gedatolisib; Drug: Paclitaxel; Drug: Carboplatin
- Treatment Arm (Phase 1b; Gedatolisib Dose Level 3[180 mg]) (Experimental)
  Interventions: Drug: Gedatolisib; Drug: Paclitaxel; Drug: Carboplatin
- Treatment Arm (Phase 2; MTD of Gedatolisib from Phase Ib) (Experimental)
  Interventions: Drug: Gedatolisib; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Gedatolisib — During the first phase, subjects will be sequentially enrolled to each increasing dose level, beginning with dose level 1 (110 mg) until the first dose limiting toxicity occurs, or safely accrued to dose level 3. PF-05212384 is intravenously infused over a thirty minute period. The dose given in the phase 2 portion will be the MTD determined in the phase Ib portion of the study.
  Dose Level 1: 110 mg Dose Level 2: 150 mg Dose Level 3: 180 mg
  Other Names: PF-05212384
Drug: Paclitaxel — Given as 200 mg/m2 infusion over a three hour period at every twenty-one days; the dose will not adjust as part of the study design.
  Other Names: Taxol®; NSC-673089
Drug: Carboplatin — The carboplatin dose (mg) = AUC x (CrCl + 25) where AUC = 6 depending on the dose level. carboplatin is intravenously infused over a thirty minute period following paclitaxel administration; the dose will not adjust as part of the study design.
  Other Names: CBDCA; NSC-241240

SUMMARY:
The purpose of this research study is to determine if the study drug, Gedatolisib (PF-05212384), given in combination with paclitaxel and carboplatin will work against unresectable non-small cell lung cancer.

DETAILED DESCRIPTION:
Approximately 70% of patients with unresectable non-small cell lung cancer (NSCLC) who receive and progress through frontline chemotherapy will be eligible for second line treatments. Any of the agents which are available for frontline therapy can be used in the salvage setting, though only erlotinib, docetaxel, and pemetrexed (in non-squamous cell carcinoma) are FDA-approved in the salvage setting based upon their demonstrated survival benefit in randomized phase III trials. All three appear to be roughly equivalent in terms of clinical benefit, which is admittedly modest, with response rates <10%, clinical benefit rates of approximately 50%, and overall survivals of approximately 6 months. Still, a substantial number of patients may not benefit from the agents in the salvage treatment setting, thus it is critical to identify those patients who stand to benefit the most.

The study will consist of two phases, Ib and II. The phase Ib portion will study dose escalations in separate 3+3 cohorts using escalating doses of PF-05212384. The phase II portion will consist of a two stage Simon design. The doses for paclitaxel (200 mg/m2, Q21 days) and carboplatin (AUC=6, Q21 days) do not adjust as part of the study design. The dose of PF-05212384 will be determined during the Phase Ib portion.

The primary endpoint of the phase Ib portion of this protocol is to determine a tolerable phase II dose of PF-05212384 in combination with paclitaxel and carboplatin. The primary endpoint of the phase II portion of this study is to determine the objective response rate of disease to the administration of PF-05212384 in combination with paclitaxel and carboplatin. A secondary endpoint of this study will be progression-free survival following PF-05212384 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed Institutional Review Board (IRB)-approved informed consent prior to any study-related procedures
* Age of 18 years or older
* Advanced-stage unresectable NSCLC, as confirmed by pathological and/or radiological analysis (subjects will be classified as having advanced disease if they were not eligible for, or had disease progression after, surgical or locoregional therapies)
* Prior chemotherapy will be allowed for other invasive malignancies, provided therapy was completed at least five years before the start of protocol therapy, and participants have recovered from all toxicities of that prior therapy
* Participants may have received prior chemotherapy for NSCLC
* In the Phase II portion, subjects must have disease which lacks PTEN expression by immunohistochemistry, or has known prior activating PI3K or inactivating PTEN gene mutations (mutations will not be assayed for specifically)
* Eastern Cooperative Oncology Group (ECOG) performance status score < 2
* Life expectancy ≥ 12 week
* Participants must have measureable disease by RECIST criteria
* Absolute neutrophil count > 1500 mm3 (individuals with benign ethnic neutropenia may be enrolled if they have no evidence of infectious diathesis, or febrile neutropenia at the time of enrollment)
* Platelet count ≥ 100×109 L
* Hgb ≥ 8.5 g/dL (subjects may receive transfusions to achieve this, in the absence of overt bleeding)
* Total Bilirubin ≤ 2 mg/dL
* aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤ 3 times the upper limit of normal range
* Serum creatinine ≤1.5 times the upper limit of the normal range
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 6 months after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal. Post-menopause is defined as:
* Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or
* For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.
* Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 6 months following the last dose of study drug

Exclusion Criteria:

* Uncontrolled cardiac disease, congestive heart failure, angina, arrhythmias or hypertension.
* Myocardial infarction or unstable angina within 2 months of treatment.
* Known human immunodeficiency virus (HIV) infection or chronic active Hepatitis B (subjects will not be screened for this).
* Active clinically serious infection > CTCAE Grade 2.
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug
* Women or men of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 6 months after the last dose of study drug
* Women who are pregnant or breastfeeding.
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects demonstrating an inability to comply with the study and/or follow-up procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennie Jones, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Cancer Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from 9/25/2017 until 12/06/2018, at which point the study was closed due to low accrual.
Groups:
- Treatment Arm (Phase 1b; Dose Level 1): Gedatolisib (Dose level 1[110 mg]), Paclitaxel, and Carboplatin
  Paclitaxel: Given as 200 mg/m2 infusion over a three hour period at every twenty-one days; the dose will not adjust as part of the study design.
  Carboplatin: The carboplatin dose (mg) = AUC x (CrCl + 25) where AUC = 6 depending on the dose level. carboplatin is intravenously infused over a thirty minute period following paclitaxel administration; the dose will not adjust as part of the study design.
- Treatment Arm (Phase 1b; Dose Level 2): Gedatolisib (Dose level 2[150 mg]), Paclitaxel, and Carboplatin
  Paclitaxel: Given as 200 mg/m2 infusion over a three hour period at every twenty-one days; the dose will not adjust as part of the study design.
  Carboplatin: The carboplatin dose (mg) = AUC x (CrCl + 25) where AUC = 6 depending on the dose level. carboplatin is intravenously infused over a thirty minute period following paclitaxel administration; the dose will not adjust as part of the study design.
- Treatment Arm (Phase 1b; Dose Level 3): Gedatolisib (Dose level 2[180 mg]), Paclitaxel, and Carboplatin
  Paclitaxel: Given as 200 mg/m2 infusion over a three hour period at every twenty-one days; the dose will not adjust as part of the study design.
  Carboplatin: The carboplatin dose (mg) = AUC x (CrCl + 25) where AUC = 6 depending on the dose level. carboplatin is intravenously infused over a thirty minute period following paclitaxel administration; the dose will not adjust as part of the study design.
- Treatment Arm (Phase 2): Gedatolisib (MTD From the Phase 1b portion), Paclitaxel, and Carboplatin
  Paclitaxel: Given as 200 mg/m2 infusion over a three hour period at every twenty-one days; the dose will not adjust as part of the study design.
  Carboplatin: The carboplatin dose (mg) = AUC x (CrCl + 25) where AUC = 6 depending on the dose level. carboplatin is intravenously infused over a thirty minute period following paclitaxel administration; the dose will not adjust as part of the study design.
Period: Overall Study
Arm/Group | Treatment Arm (Phase 1b; Dose Level 1) | Treatment Arm (Phase 1b; Dose Level 2) | Treatment Arm (Phase 1b; Dose Level 3) | Treatment Arm (Phase 2)
Started | 3 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Gedatolisib, Paclitaxel, and Carboplatin
  Gedatolisib: During the first phase, subjects will be sequentially enrolled to each increasing dose level, beginning with dose level 1 (110 mg) until the first dose limiting toxicity occurs, or safely accrued to dose level 3. PF-05212384 is intravenously infused over a thirty minute period.
  Dose Level 1: 110 mg Dose Level 2: 150 mg Dose Level 3: 180 mg
  Paclitaxel: Given as 200 mg/m2 infusion over a three hour period at every twenty-one days; the dose will not adjust as part of the study design.
  Carboplatin: The carboplatin dose (mg) = AUC x (CrCl + 25) where AUC = 6 depending on the dose level. carboplatin is intravenously infused over a thirty minute period following paclitaxel administration; the dose will not adjust as part of the study design.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose Tolerability
Description: To identify the maximum tolerated dose of PF-05212384 in combination with paclitaxel and carboplatin in subjects with NSCLC.
Time Frame: 1 year
Population: Data are not reported for this outcome measure because an insufficient number of participants were evaluable to determine the MTD.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

2. Primary Outcome: Objective Response Rate (ORR)
Description: To estimate the objective rate of response of PF-05212384 in combination with paclitaxel and carboplatin administered to subjects with unresectable or metastatic NSCLC, according to current RECIST criteria. ORR is defined as the number of participants who achieved either a partial or complete response by RECIST 1.1 criteria. By these criteria, Complete Response (CR) is defined as the disappearance of all target lesions and Partial Response (PR) is defined as a decrease of at least 30% in the sum of the longest diameter of the target lesions.
Time Frame: 1 year
Population: The sample of only 1 evaluable subject was not sufficient to analyze this outcome measure.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time a subject signed consent until 28 days after the last dose of study treatment. During this time frame, adverse event data was collected at the time informed consent was signed, on day 1 of each treatment cycle, and 28 days after the last dose of study treatment at a minimum. The time over which adverse event data was collected for the 2 subjects for whom adverse event data was collected was 2.6 and 5.75 months.
Description: Adverse events were assessed by the principal investigator, the treating sub-investigator, and/or the study coordinator from the time a subject signed consent until 28 days after the last dose of study treatment. During this time frame, adverse event data was collected at the time informed consent was signed, on day 1 of each treatment cycle, and 28 days after the last dose of study treatment at a minimum. Adverse events were assessed by physical examination, labs, and subject self-reports.
Groups:
- Treatment Arm (Phase 1b; Gedatolisib Dose Level 1[110 mg]); Treatment Arm (Phase 1b; Gedatolisib Dose Level 2[150 mg]); Treatment Arm (Phase 1b; Gedatolisib Dose Level 3[180 mg]); Treatment Arm (Phase 2; MTD of Gedatolisib From Phase Ib): Gedatolisib, Paclitaxel, and Carboplatin
  Gedatolisib: During the first phase, subjects will be sequentially enrolled to each increasing dose level, beginning with dose level 1 (110 mg) until the first dose limiting toxicity occurs, or safely accrued to dose level 3. PF-05212384 is intravenously infused over a thirty minute period.The dose given in the phase 2 portion will be the MTD determined in the phase Ib portion of the study.
  Dose Level 1: 110 mg Dose Level 2: 150 mg Dose Level 3: 180 mg
  Paclitaxel: Given as 200 mg/m2 infusion over a three hour period at every twenty-one days; the dose will not adjust as part of the study design.
  Carboplatin: The carboplatin dose (mg) = AUC x (CrCl + 25) where AUC = 6 depending on the dose level. carboplatin is intravenously infused over a thirty minute period following paclitaxel administration; the dose will not adjust as part of the study design.
Arm/Group | Treatment Arm (Phase 1b; Gedatolisib Dose Level 1[110 mg]) | Treatment Arm (Phase 1b; Gedatolisib Dose Level 2[150 mg]) | Treatment Arm (Phase 1b; Gedatolisib Dose Level 3[180 mg]) | Treatment Arm (Phase 2; MTD of Gedatolisib From Phase Ib)
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (Phase 1b; Gedatolisib Dose Level 1[110 mg]) (N=3) | Treatment Arm (Phase 1b; Gedatolisib Dose Level 2[150 mg]) (N=0) | Treatment Arm (Phase 1b; Gedatolisib Dose Level 3[180 mg]) (N=0) | Treatment Arm (Phase 2; MTD of Gedatolisib From Phase Ib) (N=0)
Sepsis (Infections and infestations) | 1 (1) | NA | NA | NA — Grade 4 Sepsis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT02920450/Prot_SAP_000.pdf